CLINICAL TRIAL: NCT05852106
Title: The Effect of 3D Modeling on Family Quality of Life, Surgical Success and Patient Outcomes in Congenital Heart Diseases: A Randomized Controlled Trial Protocol
Brief Title: The Effect of 3D Heart Modelling on Family Quality of Life and Surgical Success
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Aylin Akça, Assist Prof, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Yeditepe University Nursing
Record Dates: First submitted 2023-04-20; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart diseases; 3D printing; heart modeling; family quality of life; surgical simulation
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two hospitals affiliated with a foundation in Istanbul, located in the Marmara Region of Turkey. The imaging used in this study, including patients examined and diagnosed by the pediatric cardiology specialist doctor from the researchers involved, will be checked with a specialist radiology doctor in another hospital belonging to the same foundation. Patients included in the study will be determined with images that can be modeled and meet the inclusion and exclusion criteria. The target sample will include parents of children scheduled to undergo cardiac surgery. The study will be explained to the legal guardian/parent of the identified volunteer patients, and those who wish to participate and give written consent will be included.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Preoperative:Once the surgery date is set, appointments will be made with the surgeon for surgical simulation and with the family for education one week prior to surgery. The surgeon will be asked to complete the Surgical Simulation Evaluation Form-Part I. At the same time, another researcher will complete the family sociodemographic information form and PedsQL questions in the examination room. After completion of the pre-test and the surgical simulation, the families are given a 30-minute preoperative education with the "Congenital Heart Disease Parent Education Booklet", together with a life-size 3D heart model obtained from their child's own heart, and drawings on paper where they are not understood.
  Postoperative: After surgery, the patient will be followed until discharge, and only Part II of the Surgical Simulation Evaluation Form will be completed. On the 15th postoperative day, the Surgical Simulation Evaluation Form Part II and the PedsQL will be given again as a posttest.
  Interventions: Other: Surgical Simulation with 3D Heart Model and Parental Education with "Congenital Heart Disease Parent Education Booklet" and tailored 3D Heart Modeling
- Control Group (No Intervention): Preoperative:When the operation date is determined, one week before the operation, the patients included in the study's control group will be asked the Sociodemographic Information Form and Pediatric Quality of Life Inventory Family Module (PedQL) questions in the examination room. After the pretest, standardized education will be given to the families. The disease process will be explained to the patients with the same 'Congenital Heart Diseases Parent Education Booklet', and the disease process will be presented with the heart model used in standard medical faculty anatomy courses and the ununderstood parts will be detailed by drawing on paper. The remaining 15 minutes of the education will be conducted as a question and answer with the parents.
  Postoperative:After the operation, the Surgical Simulation Evaluation Form Part II and PedsQL will be filled out again as post-tests for this group.

INTERVENTIONS:
Other: Surgical Simulation with 3D Heart Model and Parental Education with "Congenital Heart Disease Parent Education Booklet" and tailored 3D Heart Modeling — The first step in the modeling process is masking. For this study, the average minimum value for masking ventricles and large vessels was set between 80 and 200 HU (Brüning et al., 2022). Threshold values of min 216 HU - max 1502 HU are used. At these HU values, the blood in the heart and great vessels is masked and the outline of the heart is revealed. Lowering the minimum HU value is necessary to make the heart walls more visible. However, this results in masking unwanted soft tissues other than the heart, such as muscle and fat. The masked unnecessary surrounding tissues are removed first with the cropping mask and then manually by marking along the contours of the heart and great vessels. Thus, a model containing only the heart and the desired large vessels will be created and cleaned from the surrounding tissues. With this mask, 3D reconstruction will be performed, and the model will be ready for printing.
  Other Names: Surgical Simulation with CT and MRI and Parental Education with "Congenital Heart Disease Parent Education Booklet"
  Arms: Experimental

SUMMARY:
Introduction and Objective: In recent years, 3D (three-dimensional) modeling has been added to traditional and effective diagnostic methods such as Computed Tomography (CT), Magnetic Resonance Imaging (MRI), and Echocardiography. The purpose of this study is to determine the effectiveness of models created from patients' own radiological images using 3D printing technology in the clinical setting to simulate surgery in the preoperative period and provide preoperative parental education to improve family quality of life and positively influence patient outcomes.

Methods: The study is a two-group pretest-posttest randomized controlled study. The children who come to the outpatient clinic examination in a private hospital and who are subjected to Computed Tomography (CT) examination for diagnostic procedures will be modeled in the experimental group, pre-tests will be applied, and the model will be 3D printed after it is approved by the radiologist who is among the researchers. The sample size is 15 experimental group and 15 control group. After the radiologist's approval, surgical simulation and preoperative education will be applied to the experimental group. The control group will receive the same parent education as the standard model. Both groups will complete the Sociodemographic Information Form, Surgical Simulation Evaluation Form - Part I, and Pediatric Quality of Life Inventory (PedsQL) Family Impacts Module one week prior to hospitalization. Surgical simulation and preoperative education will be completed on the same day. On postoperative day 0, only the Surgical Simulation Evaluation Form - Part II will be applied and on postoperative day 15, the Surgical Simulation Evaluation Form - Part II and the Pediatric Quality of Life Inventory (PedsQL) Family Impacts Module will be applied to both groups as a posttest.

Pilot Study and Results: Modeling and 3D printing studies were conducted to carry out the study. A total of four diagnosed and treated patients were retrospectively analyzed. An intracardiac anomaly was detected in the patient data taken for the first model. It was decided to model the extracardiac structures since the inside of the heart was filled with blood, and the blood could not be ruled out as a solid structure. Finally, aortic coarctation was modeled clearly from the images taken and completed.

DETAILED DESCRIPTION:
The most common congenital malformation of childhood is congenital heart disease (CHD). The degree to which the defect deviates from normal anatomy determines the severity of symptoms. Globally, between 0.8% and 1.2% of all live births are affected by CHD. While it occurs in 1% of 40,000 live births in the US, Asian countries have been reported to have the highest rate at 9.3 per 1000 live births. In Turkey, the rate has been reported to be between 0.6 and 1% per 100 live births. Between 25 % and 50 % of the children born with CHD have defects that will require open heart surgery. Reliable diagnostic methods provide much better treatment options, leading to a significant reduction in mortality. In addition to imaging methods such as Computed Tomography (CT), Magnetic Resonance Imaging (MRI), and Echocardiography (ECHO), 3D modeling and printing technologies have been added to these methods in recent years. There are differences and benefits among the different imaging methods. The most recent and rapidly developing method among them is 3D printing technologies.

It is predicted that 3D cardiac models obtained from patients' radiological images can be used for various purposes. It is stated that beneficial results can be obtained for multiple purposes, from planning and simulation before the definitive surgical procedure to patient-specific preoperative education. There are several techniques for modeling organs using 3D printing technology, which has developed rapidly in recent years. For the heart, two types of cardiac modeling are performed. These are filled solid models (blood pool) and hollow models. The hollow models are obtained from signals sent in a way that limits the perimeter of the area where the blood pool is located. These models are printed as a cross-section and show the intracardiac structure. However, technically, the peak heart rate of children is higher than that of adults, so the images may lose clarity, require more time and effort, and may not be as useful. Solid models have filled models of the atria and ventricles. They are typically modeled and printed from contrast-enhanced CT or MR images. Noncardiac structures can be added to these models (e.g., aorta, pulmonary artery, extracardiac vessels, trachea, and esophagus) with the goal of delineating large vessel abnormalities in the model. Extracardiac structures are very guiding in surgical simulation with easier and faster modeling than intracardiac structures. In particular, recurrent pulmonary artery stenosis and aortic coarctation can be successfully treated, and positive outcomes can be achieved with fast and patient-specific models. The operating time of surgically simulated patients is reduced, and procedures can be completed with less cost and fewer complications.

Targeted patient outcomes can be achieved by managing a multidisciplinary team that includes the patient and family and by using surgical simulation. In life-threatening diseases such as CHD, diagnosis, treatment, and surgical planning are long-term processes. This process causes serious psychological distress in parents, such as post-traumatic stress disorder. Parental/caregiver stress increases and the family's quality of life deteriorates, especially when the surgical procedure and interventions are not clearly understood. This situation negatively affects the postoperative recovery process of patients. A surgical procedure performed with good technique followed by poor postoperative management renders many interventions ineffective. Understanding the severity of the disease from the perspective of the parents can improve both the health-related quality of life of the child and the quality of life of the family, leading to more positive patient outcomes. Patient-specific modeling using 3D printing technology with images obtained through traditional methods is believed to eliminate all of these issues.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a congenital heart disease between the ages of 0-18 years, the congenital defect has extracardiac structure malformations (This is because the modeling is to be done before the operation is done in a shorter time, and it is desired to be trained for preoperative education). Hollow modeling requires more detailed technique and time (Bhatla et al., 2017). In addition, the difficulty of 3D printing the hollow model made in the pilot study was also effective in this decision),
* Being a candidate for elective surgery,
* Having a contrast-enhanced CT image taken during and before the patient's routine diagnostic procedure outside the scope of the study,
* Having at least 15 days between the imaging and the surgical procedure plan,
* The parents/legal guardians who gave permission to participate in the study were the inclusion criteria of the study.

Exclusion Criteria:

* Patients who do not require CT for diagnosis or treatment (no patient will undergo CT imaging within the scope of the study unless necessary for this study only),
* Emergency surgical procedures, heart defects involving intracardiac structures (Atrial Septal Defect, Ventricular Septal Defect, Tetralogy of Fallot),
* Additional anomalies/syndromes,
* Chronic diseases (such as neurodevelopmental disorders, bleeding disorders, asthma, or Down syndrome),
* History of cardiac arrest, contrast agent reflection in the images,
* Image quality preventing modeling.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pretest-Family Impacts Module of the Pediatric Quality of Life Inventory PedsQL | 1 week prior to surgery
  The Turkish validity and reliability study of this scale, first developed by Varni et al. in 2004, was conducted and published by Gürkan et al. in 2019 (Gürkan, Bahar, Çapık, Aydoğdu, & Beşer, 2020; Varni, Sherman, Burwinkle, Dickinson, & Dixon, 2004). The data on the sub-dimensions and Cronbach alpha values of this scale, which has 8 sub-dimensions in total, are as follows; physical (0.85), emotional (0.83), social (0.82), cognitive (0.86), communication (0.51), anxiety (0.79) activities of daily living (0.89), family relationships (0.95). A total score of 0.92 was reported. In addition, Cronbach alpha values for all subscales were also included in the original study. The scale does not have a cut-off point. A high score indicates a good family quality of life functioning, while a low score indicates a negative family quality of life. Within the scope of this study, a comparison between mean scores will be made.
Posttest-Family Impacts Module of the Pediatric Quality of Life Inventory PedsQL | 15 days later to surgery
  The Turkish validity and reliability study of this scale, first developed by Varni et al. in 2004, was conducted and published by Gürkan et al. in 2019 (Gürkan, Bahar, Çapık, Aydoğdu, & Beşer, 2020; Varni, Sherman, Burwinkle, Dickinson, & Dixon, 2004). The data on the sub-dimensions and Cronbach alpha values of this scale, which has 8 sub-dimensions in total, are as follows; physical (0.85), emotional (0.83), social (0.82), cognitive (0.86), communication (0.51), anxiety (0.79) activities of daily living (0.89), family relationships (0.95). A total score of 0.92 was reported. In addition, Cronbach alpha values for all subscales were also included in the original study. The scale does not have a cut-off point. A high score indicates a good family quality of life functioning, while a low score indicates a negative family quality of life. Within the scope of this study, a comparison between mean scores will be made.
Posttest-Surgical Simulation Questionnaire Part II | First post operative day
  It has 7 questions prepared according the literature. Effects of 3D modeling on surgical complications, duration of the operation, duration of the hospitalization, duration of the intensive care unit, need of recurrent surgery, Unusual complications (except for pain, cardiopulmonary resuscitation, need for ECMO (Extracorporeal Membrane Oxygenation), Seizure, rhythm changes, etc.)
Posttest-Surgical Simulation Questionnaire Part II | 15 days later to surgery
  It has 7 questions prepared according the literature. Effects of 3D modeling on surgical complications, duration of the operation, duration of the hospitalization, duration of the intensive care unit, need of recurrent surgery, Unusual complications (except for pain, cardiopulmonary resuscitation, need for ECMO (Extracorporeal Membrane Oxygenation), Seizure, rhythm changes, etc.)

SECONDARY OUTCOMES:
Pretest Surgical Simulation Questionnaire Part I | 1 week prior to surgery
  Surgeon's professional experience and age, opinions about 3D Heart Modeling (surgical simulation evaluations such as effectiveness on techniques of the operations, opinions about strong and week sides of 3D modeling)

CONTACTS AND LOCATIONS:
Overall Officials: AYLIN AKCA SUMENGEN, PhD, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Researchers will ensure that all data are accurately and completely coded and consistently entered into the statistical analysis software. The researchers will keep all original documents including medical records, questionnaires, informed consent forms, and other relevant records obtained during the study and will keep them confidential. Data will be retained for five years after the completion of the study.

REFERENCES:
- [Background] Abdullah KA, Reed W. 3D printing in medical imaging and healthcare services. J Med Radiat Sci. 2018 Sep;65(3):237-239. doi: 10.1002/jmrs.292. Epub 2018 Jul 3. PMID 29971971
- [Background] AHA. (2023). How 3D Printing Is Impacting Clinical Care. Anatomical Models. Retrieved from https://www.aha.org/aha-center-health-innovation-market-scan/2022-06-07-3-ways-3d-printing-revolutionizing-health-care
- [Background] Anwar S, Singh GK, Miller J, Sharma M, Manning P, Billadello JJ, Eghtesady P, Woodard PK. 3D Printing is a Transformative Technology in Congenital Heart Disease. JACC Basic Transl Sci. 2018 May 30;3(2):294-312. doi: 10.1016/j.jacbts.2017.10.003. eCollection 2018 Apr. PMID 30062215
- [Background] Atalay, B., Güler, R., & Haylı, Ç. M. (2021). Investigation of Preoperative Anxiety Levels in Pediatric Groups. Turkish Journal of Health Science and Life, 4(1), 24-26.
- [Background] Awori J, Friedman SD, Chan T, Howard C, Seslar S, Soriano BD, Buddhe S. 3D models improve understanding of congenital heart disease. 3D Print Med. 2021 Sep 2;7(1):26. doi: 10.1186/s41205-021-00115-7. PMID 34471999
- [Background] Azhar AS, AlShammasi ZH, Higgi RE. The impact of congenital heart diseases on the quality of life of patients and their families in Saudi Arabia. Biological, psychological, and social dimensions. Saudi Med J. 2016 Apr;37(4):392-402. doi: 10.15537/smj.2016.4.13626. PMID 27052282
- [Background] Ballard DH, Mills P, Duszak R Jr, Weisman JA, Rybicki FJ, Woodard PK. Medical 3D Printing Cost-Savings in Orthopedic and Maxillofacial Surgery: Cost Analysis of Operating Room Time Saved with 3D Printed Anatomic Models and Surgical Guides. Acad Radiol. 2020 Aug;27(8):1103-1113. doi: 10.1016/j.acra.2019.08.011. Epub 2019 Sep 18. PMID 31542197
- [Background] Barsella, R. (2020). Pilot Study: Educational Tool Reduces Parental Stress at Home Post Pediatric Cardiac Surgery.
- [Background] Bhatla P, Tretter JT, Ludomirsky A, Argilla M, Latson LA Jr, Chakravarti S, Barker PC, Yoo SJ, McElhinney DB, Wake N, Mosca RS. Utility and Scope of Rapid Prototyping in Patients with Complex Muscular Ventricular Septal Defects or Double-Outlet Right Ventricle: Does it Alter Management Decisions? Pediatr Cardiol. 2017 Jan;38(1):103-114. doi: 10.1007/s00246-016-1489-1. Epub 2016 Nov 11. PMID 27837304
- [Background] Bibb, R., Eggbeer, D., & Paterson, A. (2014). Medical modelling: the application of advanced design and rapid prototyping techniques in medicine: Woodhead Publishing.
- [Background] Biber S, Andonian C, Beckmann J, Ewert P, Freilinger S, Nagdyman N, Kaemmerer H, Oberhoffer R, Pieper L, Neidenbach RC. Current research status on the psychological situation of parents of children with congenital heart disease. Cardiovasc Diagn Ther. 2019 Oct;9(Suppl 2):S369-S376. doi: 10.21037/cdt.2019.07.07. PMID 31737543
- [Background] Bouma BJ, Mulder BJ. Changing Landscape of Congenital Heart Disease. Circ Res. 2017 Mar 17;120(6):908-922. doi: 10.1161/CIRCRESAHA.116.309302. PMID 28302739
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Boyer PJ, Yell JA, Andrews JG, Seckeler MD. Anxiety reduction after pre-procedure meetings in patients with CHD. Cardiol Young. 2020 Jul;30(7):991-994. doi: 10.1017/S1047951120001407. Epub 2020 Jun 5. PMID 32500844
- [Background] Bruning J, Kramer P, Goubergrits L, Schulz A, Murin P, Solowjowa N, Kuehne T, Berger F, Photiadis J, Weixler VH. 3D modeling and printing for complex biventricular repair of double outlet right ventricle. Front Cardiovasc Med. 2022 Nov 30;9:1024053. doi: 10.3389/fcvm.2022.1024053. eCollection 2022. PMID 36531701
- [Background] Burkhart HM. Simulation in congenital cardiac surgical education: We have arrived. J Thorac Cardiovasc Surg. 2017 Jun;153(6):1528-1529. doi: 10.1016/j.jtcvs.2017.03.012. Epub 2017 Mar 10. No abstract available. PMID 28359578
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Chaudhuri, A., Naseraldin, H., Soberg, P. V., Kroll, E., & Librus, M. (2020). Should hospitals invest in customised on-demand 3D printing for surgeries? International Journal of Operations & Production Management, 41(1), 55-62.
- [Background] Çil, E. (2006). Konjenital kalp hastalıkları. Turkiye Klinikleri J Int Med Sci, 2(15), 51-59.
- [Background] Farooqi, K. M. (2017). Rapid prototyping in cardiac disease: Springer.
- [Background] Feins RH. Expert commentary: Cardiothoracic surgical simulation. J Thorac Cardiovasc Surg. 2008 Mar;135(3):485-6. doi: 10.1016/j.jtcvs.2008.01.001. No abstract available. PMID 18329456
- [Background] Gürkan, K. P., Bahar, Z., Çapık, C., Aydoğdu, N. G., & Beşer, A. (2020). Psychometric properties of the Turkish version of the pediatric quality of life: The family impact module in parents of children with type 1 diabetes. Children's Health Care, 49(1), 87-99.
- [Background] Hartman DM, Medoff-Cooper B. Transition to home after neonatal surgery for congenital heart disease. MCN Am J Matern Child Nurs. 2012 Mar-Apr;37(2):95-100. doi: 10.1097/NMC.0b013e318241dac1. PMID 22357070
- [Background] Hounsfield GN. Computed medical imaging. Nobel lecture, Decemberr 8, 1979. J Comput Assist Tomogr. 1980 Oct;4(5):665-74. doi: 10.1097/00004728-198010000-00017. No abstract available. PMID 6997341
- [Background] Kain A, Mueller C, Golianu BJ, Jenkins BN, Fortier MA. The impact of parental health mindset on postoperative recovery in children. Paediatr Anaesth. 2021 Mar;31(3):298-308. doi: 10.1111/pan.14071. Epub 2020 Nov 29. PMID 33187011
- [Background] Ladak LA, Hasan BS, Gullick J, Awais K, Abdullah A, Gallagher R. Health-related quality of life in surgical children and adolescents with congenital heart disease compared with their age-matched healthy sibling: a cross-sectional study from a lower middle-income country, Pakistan. Arch Dis Child. 2019 May;104(5):419-425. doi: 10.1136/archdischild-2018-315594. Epub 2018 Dec 15. PMID 30554150
- [Background] Lau IWW, Liu D, Xu L, Fan Z, Sun Z. Clinical value of patient-specific three-dimensional printing of congenital heart disease: Quantitative and qualitative assessments. PLoS One. 2018 Mar 21;13(3):e0194333. doi: 10.1371/journal.pone.0194333. eCollection 2018. PMID 29561912
- [Background] Liddle D, Balsara S, Hamann K, Christopher A, Olivieri L, Loke YH. Combining patient-specific, digital 3D models with tele-education for adolescents with CHD. Cardiol Young. 2022 Jun;32(6):912-917. doi: 10.1017/S1047951121003243. Epub 2021 Aug 16. PMID 34392874
- [Background] Liu Y, Chen S, Zuhlke L, Black GC, Choy MK, Li N, Keavney BD. Global birth prevalence of congenital heart defects 1970-2017: updated systematic review and meta-analysis of 260 studies. Int J Epidemiol. 2019 Apr 1;48(2):455-463. doi: 10.1093/ije/dyz009. PMID 30783674
- [Background] Lopez, C., Hanson, C. C., Yorke, D., Johnson, J. K., Mill, M. R., Brown, K. J., & Barach, P. (2017). Improving communication with families of patients undergoing pediatric cardiac surgery. Progress in Pediatric Cardiology, 45, 83-90.
- [Background] Mahesh M. Search for isotropic resolution in CT from conventional through multiple-row detector. Radiographics. 2002 Jul-Aug;22(4):949-62. doi: 10.1148/radiographics.22.4.g02jl14949. PMID 12110725
- [Background] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541
- [Background] Ngan EM, Rebeyka IM, Ross DB, Hirji M, Wolfaardt JF, Seelaus R, Grosvenor A, Noga ML. The rapid prototyping of anatomic models in pulmonary atresia. J Thorac Cardiovasc Surg. 2006 Aug;132(2):264-9. doi: 10.1016/j.jtcvs.2006.02.047. PMID 16872948
- [Background] Olivieri LJ, Su L, Hynes CF, Krieger A, Alfares FA, Ramakrishnan K, Zurakowski D, Marshall MB, Kim PC, Jonas RA, Nath DS. "Just-In-Time" Simulation Training Using 3-D Printed Cardiac Models After Congenital Cardiac Surgery. World J Pediatr Congenit Heart Surg. 2016 Mar;7(2):164-8. doi: 10.1177/2150135115623961. PMID 26957398
- [Background] Puranik R, Muthurangu V, Celermajer DS, Taylor AM. Congenital heart disease and multi-modality imaging. Heart Lung Circ. 2010 Mar;19(3):133-44. doi: 10.1016/j.hlc.2010.01.001. Epub 2010 Feb 23. PMID 20181524
- [Background] Raju TN. The Nobel chronicles. 1979: Allan MacLeod Cormack (b 1924); and Sir Godfrey Newbold Hounsfield (b 1919). Lancet. 1999 Nov 6;354(9190):1653. doi: 10.1016/s0140-6736(05)77147-6. No abstract available. PMID 10560712
- [Background] Ruggiero KM, Hickey PA, Leger RR, Vessey JA, Hayman LL. Parental perceptions of disease-severity and health-related quality of life in school-age children with congenital heart disease. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12204. Epub 2017 Dec 20. PMID 29266743
- [Background] Ryan JR, Moe TG, Richardson R, Frakes DH, Nigro JJ, Pophal S. A novel approach to neonatal management of tetralogy of Fallot, with pulmonary atresia, and multiple aortopulmonary collaterals. JACC Cardiovasc Imaging. 2015 Jan;8(1):103-104. doi: 10.1016/j.jcmg.2014.04.030. Epub 2014 Nov 12. No abstract available. PMID 25457761
- [Background] Shiraishi I, Yamagishi M, Hamaoka K, Fukuzawa M, Yagihara T. Simulative operation on congenital heart disease using rubber-like urethane stereolithographic biomodels based on 3D datasets of multislice computed tomography. Eur J Cardiothorac Surg. 2010 Feb;37(2):302-6. doi: 10.1016/j.ejcts.2009.07.046. Epub 2009 Sep 15. PMID 19758813
- [Background] Simeone S, Platone N, Perrone M, Marras V, Pucciarelli G, Benedetti M, Dell'Angelo G, Rea T, Guillari A, Da Valle P, Gargiulo G, Botti S, Artioli G, Comentale G, Ferrigno S, Palma G, Baratta S. The lived experience of parents whose children discharged to home after cardiac surgery for congenital heart disease. Acta Biomed. 2018 Apr 4;89(4-S):71-77. doi: 10.23750/abm.v89i4-S.7223. PMID 29644992
- [Background] Staveski SL, Boulanger K, Erman L, Lin L, Almgren C, Journel C, Roth SJ, Golianu B. The Impact of Massage and Reading on Children's Pain and Anxiety After Cardiovascular Surgery: A Pilot Study. Pediatr Crit Care Med. 2018 Aug;19(8):725-732. doi: 10.1097/PCC.0000000000001615. PMID 29912070
- [Background] Tabachnick, B., & Fidell, L. (2014). Pearson new international edition: Using multivariate statistics (Sixth). In: Pearson Education Limited
- [Background] Tack P, Willems R, Annemans L. An early health technology assessment of 3D anatomic models in pediatric congenital heart surgery: potential cost-effectiveness and decision uncertainty. Expert Rev Pharmacoecon Outcomes Res. 2021 Oct;21(5):1107-1115. doi: 10.1080/14737167.2021.1879645. Epub 2021 Feb 20. PMID 33475446
- [Background] Tenhoff, A. C., Aggarwal, V., Ameduri, R., Deakyne, A., Iles, T. L., Said, S. M., . . . Iaizzo, P. A. (2021). Patient-Specific Three-Dimensional Computational Heart Modeling and Printing to Enhance Clinical Understandings and Treatment Planning: Congenital Recurrent Pulmonary Artery Stenosis and Transcatheter Pulmonary Valve Replacement. Paper presented at the 2021 Design of Medical Devices Conference.
- [Background] Valverde I, Gomez-Ciriza G, Hussain T, Suarez-Mejias C, Velasco-Forte MN, Byrne N, Ordonez A, Gonzalez-Calle A, Anderson D, Hazekamp MG, Roest AAW, Rivas-Gonzalez J, Uribe S, El-Rassi I, Simpson J, Miller O, Ruiz E, Zabala I, Mendez A, Manso B, Gallego P, Prada F, Cantinotti M, Ait-Ali L, Merino C, Parry A, Poirier N, Greil G, Razavi R, Gomez-Cia T, Hosseinpour AR. Three-dimensional printed models for surgical planning of complex congenital heart defects: an international multicentre study. Eur J Cardiothorac Surg. 2017 Dec 1;52(6):1139-1148. doi: 10.1093/ejcts/ezx208. PMID 28977423
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432
- [Background] Varni JW, Sherman SA, Burwinkle TM, Dickinson PE, Dixon P. The PedsQL Family Impact Module: preliminary reliability and validity. Health Qual Life Outcomes. 2004 Sep 27;2:55. doi: 10.1186/1477-7525-2-55. PMID 15450120
- [Background] Wang AT, Sundt TM 3rd, Cutshall SM, Bauer BA. Massage therapy after cardiac surgery. Semin Thorac Cardiovasc Surg. 2010 Autumn;22(3):225-9. doi: 10.1053/j.semtcvs.2010.10.005. PMID 21167456
- [Background] Wu W, He J, Shao X. Incidence and mortality trend of congenital heart disease at the global, regional, and national level, 1990-2017. Medicine (Baltimore). 2020 Jun 5;99(23):e20593. doi: 10.1097/MD.0000000000020593. PMID 32502030
- [Background] Yoo SJ, Spray T, Austin EH 3rd, Yun TJ, van Arsdell GS. Hands-on surgical training of congenital heart surgery using 3-dimensional print models. J Thorac Cardiovasc Surg. 2017 Jun;153(6):1530-1540. doi: 10.1016/j.jtcvs.2016.12.054. Epub 2017 Feb 9. PMID 28268011
- [Background] Yoo SJ, Hussein N, Peel B, Coles J, van Arsdell GS, Honjo O, Haller C, Lam CZ, Seed M, Barron D. 3D Modeling and Printing in Congenital Heart Surgery: Entering the Stage of Maturation. Front Pediatr. 2021 Feb 5;9:621672. doi: 10.3389/fped.2021.621672. eCollection 2021. PMID 33614554